CLINICAL TRIAL: NCT05075655
Title: Diagnosis of Lymphoma Using Endobronchial Ultrasound Guided Miniforceps Biopsy.
Brief Title: Endobronchial Diagnosis of Lymphoma
Acronym: EnDol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-028
Record Dates: First submitted 2021-09-15; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Lymphoma
Keywords: ebus; endobronchial ultrasound-guided; EBUS-MFB; intra-nodal miniforceps biopsy; EBUS-transbronchial forceps biopsy
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Masking Description: pathologist do not know the technique of sampling used when analysing slides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBUS-MFB and EBUS-TBNA (Experimental): patient will have both TBNA and MFB in the same operating time
  Interventions: Device: Endobronchial ultrasound guided miniforceps biopsy and transbronchial needle aspiration

INTERVENTIONS:
Device: Endobronchial ultrasound guided miniforceps biopsy and transbronchial needle aspiration — Mediastinal node is sampled using three path of classic ultrasound guided transbronchial needle aspiration (EBUS-TBNA).
  A reduce size forceps is then inserted inside the mediastinal node via the duc EBUS-TBNA made and biopsies (EBUS-MFB) are made using real time ultrasound guidance.

SUMMARY:
The present study aimed to assess the diagnostic performance of ultrasound-guided endobronchial intra-nodal miniforceps biopsy (EBUS-MFB) in the diagnosis of "de novo" mediastinal lymphoma.

DETAILED DESCRIPTION:
Every patients will be sampled using both EBUS-MFB and the standard of care EBUS-TBNA (transbronchial needle aspiration).

It is a monocentric investigation. Pathologist will not know the way of sampling while analysing the samples

ELIGIBILITY:
Inclusion Criteria:

* Pathological mediastinal nodes within reach of EBUS sampling on CT-scan.
* Lymphoma suspicion by a senior clinical hematologist
* Affiliated to the french public health care insurance

Exclusion Criteria:

* Peripherical pathological lymph nodes reachable without general anesthesia
* Antithrombotic medication that cannot be stopped le time of the procedure.
* Unstable respiratory status
* History of lymphoma
* Latex or xylocaine allergia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
positivity of the procedure in Diagnosis and Subtyping of lymphoma | up to 3 years
  a sample wil be considered positive if it allows the clinical management of the patient, without additional sampling required.

SECONDARY OUTCOMES:
every adverse effect related to the procedure | up to 3 years
  infectious process related to the procedure, hemoptysis over 50cc, worsening of respiratory status requiring hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- CaenUH, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No